CLINICAL TRIAL: NCT00746213
Title: Chronic Pain After Thoracotomy, an Incidence Study
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Lung Cancer Group (Other); Aarhus University Hospital (Other)
Responsible Party: MD, Kim Wildgaard, Section for Surgical Pathophysiology 4074
Other Study IDs: H-B-2008-059; 2007-58-0015
Record Dates: First submitted 2008-07-30; First posted 2008-09-03 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Thoracotomy; Chronic Pain
Keywords: Thoracotomy; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an investigation on the frequency of chronic pain after thoracotomy for lung cancer. Factors relating to the development of chronic pain are investigated. Questionnaire survey.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give consent
* Can read
* Residing in Denmark

Exclusion Criteria:

* Unable to understand the written information in Danish
* Abuse (Medicine, Drugs, Alcohol)
* Severe psychiatric Illness
* Conflicting neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post thoracotomy patients after lung cancer in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 1340 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Pain and pain score | more than 6 months postoperative

SECONDARY OUTCOMES:
Activity of daily life | >6 months
Analgesic consumption and pain treatment | >6 months

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, MD.Phd,Proff, Study Chair — Section for Surgical Pathophysiology 4074
Locations (1):
- Section for Surgical Pathophysiology 4074, Copenhagen, Denmark